CLINICAL TRIAL: NCT04256967
Title: Body Appearance Pressure and Body Image Among University Students
Brief Title: Body Image Among University Students
Status: Completed | Type: Observational
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: University College of Southeast Norway (Other); University of Agder (Other); Ostfold University College (Other)
Responsible Party: Principal Investigator, Professor Jorunn Sundgot-Borgen, Professor, Norwegian School of Sport Sciences
Other Study IDs: CSB
Record Dates: First submitted 2020-01-11; First posted 2020-02-05 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2022-04

CONDITIONS: Body Image; Body Image Disturbance; Physical Activity; Dietary Habits; Quality of Life
MeSH Terms: conditions — Motor Activity; Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sport sciences: Bachelor and master students who study sport science or physical activity and health science
  Interventions: Other: Body and health focused study environment
- Controls: Bachelor and master students who study other fields not related to sport or physical activity and health sciences.

INTERVENTIONS:
Other: Body and health focused study environment — Students are exposed to lectures, literature, co-students, contexts that provide body and lifestyle awareness beyond the existing exposure of the society in general
  Groups: Sport sciences

SUMMARY:
A negative body image negatively affects the total health of students and the quality of life in University students. Body image and the experience of body appearance pressure have not been investigated previously among the Norwegian student population. It is reasonable to suggest that sport science students experience an increased pressure to have an athletic body to be able to identify as a sport science student and for future job opportunities. Such pressure would negatively influence students' attitudes and practice as future communicators of lifestyle knowledge after completing their studies. Objective: The study objective is to assess body image and body appearance pressure among Norwegian University students, and to investigate differences between different academic disciplines and gender. The study uses a cross-sectional design with a questionnaire to measure outcomes in male and female students in Norway.

DETAILED DESCRIPTION:
Background: A negative body image negatively affects the total health of students and the quality of life in University students. Body image and the experience of body appearance pressure have not been investigated previously among the Norwegian student population. It is well known that students studying sport science are exposed to an enhanced focus on lifestyle and the body beyond what focus that already exist in the society. It is reasonable to suggest that sport science students experience an increased pressure to have an athletic body to be able to identify as a sport science student and for future job opportunities. Such pressure would negatively influence students' attitudes and practice as future communicators of lifestyle knowledge after completing their studies. Objective: The study objective is to assess body image and body appearance pressure among Norwegian University students, and to investigate differences between different academic disciplines and gender. Methods:

The study uses a cross-sectional design with a web-based questionnaire to measure outcomes in 1764 male and female students in Norway. In addition to descriptive data on the sample, a Pearson's correlation, independent t-test og chi-square will be used to investigate associations and differences between groups. Statistical significance is defined at a p-value of <.05. Implications: Results from the study provides a description of the sample and will provide a foundation for targeted actions, interventions for optimization in terms of study environment to reduce negative body image and potential reported pressure to have a specific body, and promotion of positive body image and prevention of negative body experiences. This could contribute to a healthier student environment and enhances the chance to develop students who adapts and take knowledge with them into their future work life, and apply this knowledge in a safe and health promotive way.

ELIGIBILITY:
Inclusion Criteria:

* Students at Norwegian University Colleges or Universities
* Students who are able to read and write in Norwegian
* Fulltime students

Exclusion Criteria:

* Students who are not able to read or write in Norwegian
* Part-time students

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The sample represents students at University Colleges and Universities located in the south, east, west, and north of Norway. Both students in a sport science or physical activity and health science study program, and students who follow non-sport science study programs are represented.
Sampling Method: Non-Probability Sample
Enrollment: 993 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Self-developed | March 2020-July 2020
  Body appearance pressure. Respond on a Likert-scale where higher scores indicate higher level of experienced pressure
Body Appreciation Scale-2 | March 2020-July 2020
  Positive body image. Score ranges from 10-50, with higher score indicating higher body appreciation.
Eating Disorder Examination-Questionnaire (EDE-Q) | March 2020-July 2020
  Body dissatisfaction in girls. Scores ranges from 12-60, with higher scores indicating higher levels of dissatisfaction
Male body dissatisfaction scale (MBDS) | March 2020-July 2020
  Body dissatisfaction in males. Scores ranges from 0-42, with higher scores indicating higher levels of dissatisfaction

OTHER OUTCOMES:
Physical Appearance Comparison Scale-Revised (PACS-R) | March 2020-July 2020
  Comparison of physical appearance. Scores ranges from 0-44, where higher score indicates higher level of comparison.
Social attitudes towards appearance questionnaire (SATAQ-4 R) men | March 2020-July 2020
  Body ideal internalization. Scores ranged from 8-40, with higher score indicating higher level of internalization
Social attitudes towards appearance questionnaire (SATAQ-4 R) women | March 2020-July 2020
  Body ideal internalization. Scores ranged from 15-75, with higher score indicating higher level of internalization
Rosenberg self-esteem scale | March 2020-July 2020
  Self-esteem. Scale ranges from 10-40, with higher scores indicating higher level of self-esteem
  Self-esteem. The scale ranges from 10-40, with higher score indicates higher level of self-esteem
Satisfaction with Life Scale (SWLS) | March 2020-July 2020
  Satisfaction with life. Scores ranges from 10-70, with higher score indicating higher satisfaction with life
Physical activity level | March 2020-July 2020
  Questions about hours of physical activity during one regular week. Continuous scale.
Dietary supplementation consumption | March 2020-July 2020
  Questions about the use of dietary supplementation, both legal and illegal. Responds is given by choosing specific supplementations

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn Sundgot-Borgen, PhD, Principal Investigator — The Norwegian School of Sport Sciences
Locations (1):
- Norwegian school of sport sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Unidentifiable data can be shared between researcher within the research group.

REFERENCES:
- [Result] Sundgot-Borgen C, Sundgot-Borgen J, Bratland-Sanda S, Kolle E, Torstveit MK, Svantorp-Tveiten KME, Mathisen TF. Body appreciation and body appearance pressure in Norwegian university students comparing exercise science students and other students. BMC Public Health. 2021 Mar 19;21(1):532. doi: 10.1186/s12889-021-10550-0. PMID 33740918
- [Result] Sundgot-Borgen C, Mathisen TF, Torstveit MK, Sundgot-Borgen J. Explanations for use of dietary- and muscle enhancing dietary supplements among university students: a national cross-sectional study. BMC Nutr. 2022 Feb 24;8(1):17. doi: 10.1186/s40795-022-00510-1. PMID 35209960